CLINICAL TRIAL: NCT02629861
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study Comparing the Efficacy and Safety of 2 Dose Regimens of Subcutaneous Administration of Fremanezumab (TEV-48125) vs Placebo for the Preventive Treatment of Episodic Migraine
Brief Title: Efficacy and Safety of 2 Dose Regimens of TEV-48125 Versus Placebo for the Preventive Treatment of Episodic Migraine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TV48125-CNS-30050; 2015-004598-34 (EudraCT Number)
Record Dates: First submitted 2015-12-10; First posted 2015-12-14 (Estimated); Results first posted 2018-11-08 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — fremanezumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Matching Placebo
  Interventions: Drug: Placebo
- Fremanezumab 675 mg/placebo/placebo (Experimental): Participants randomized to receive fremanezumab 675 mg/placebo/placebo received 675 mg of fremanezumab as 3 injections (225 mg/1.5 mL) on Day 0, and placebo as a single 1.5-mL injection on Days 28 and 56.
  Interventions: Drug: Fremanezumab; Drug: Placebo
- Fremanezumab 225/225/225 mg (Experimental): Participants randomized to receive fremanezumab 225/225/225 mg received 1 active injection (225 mg/1.5 mL) on Days 0, 28 and 56.
  Interventions: Drug: Fremanezumab

INTERVENTIONS:
Drug: Fremanezumab — Fremanezumab was provided as a sterile, unpreserved, aqueous solution for injection, 225 mg/1.5 mL pre-filled syringe for single-use administration.
  The 675 mg dose was given as 3 injections; doses of 225 mg were given as a single injection. Study drug was administered at the clinical site.
  Other Names: TEV-48125, anti-calcitonin gene-related peptide (anti-CGRP)
  Arms: Fremanezumab 225/225/225 mg; Fremanezumab 675 mg/placebo/placebo
Drug: Placebo — Placebo 1.5 mL pre-filled syringes identical in appearance to active intervention. Study drug was administered at the clinical site.
  Arms: Fremanezumab 675 mg/placebo/placebo; Placebo

SUMMARY:
The study is being conducted to evaluate two doses of TEV-48125 in adult patients with episodic migraine

ELIGIBILITY:
Inclusion Criteria:

* Males or females aged 18 to 70 years, inclusive, with migraine onset at ≤50 years of age
* Patient signs and dates the informed consent document
* Patient has history of migraine according to International Classification of Headache Disorders, or clinical judgment suggests a migraine diagnosis
* 85% e-diary compliance
* Total body weight between 99 and 265 lbs, inclusive

  * Additional criteria apply, please contact the investigator for more information

Exclusion Criteria:

* Clinically significant hematological, cardiac, renal, endocrine, pulmonary, gastrointestinal, genitourinary, neurologic, hepatic, or ocular disease, at the discretion of the investigator
* Evidence or medical history of clinically significant psychiatric issues, including any suicide attempt in the past, or suicidal ideation with a specific plan in the past 2 years
* History of clinically significant cardiovascular disease or vascular ischemia (such as myocardial, neurological [eg, cerebral ischemia], peripheral extremity ischemia, or other ischemic event) or thromboembolic events (arterial or venous thrombotic or embolic events), such as cerebrovascular accident (including transient ischemic attacks), deep vein thrombosis, or pulmonary embolism
* Known infection or history of human immunodeficiency virus, tuberculosis, or chronic hepatitis B or C infection
* Past or current history of cancer in the last 5 years, except for appropriately treated nonmelanoma skin carcinoma
* Pregnant or nursing females
* History of hypersensitivity reactions to injected proteins, including monoclonal antibodies
* Participation in a clinical study of a new chemical entity or a prescription medicine within 2 months or 5 half-lives, whichever is longer

  * Additional criteria apply, please contact the investigator for more information

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 875 (Actual)
Dates: Start 2016-03-23 (Actual); Primary Completion 2017-04-10 (Actual); Study Completion 2017-04-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teva Medical Expert, MD, Study Director — Teva Branded Pharmaceutical Products R&D, Inc.
Locations (150):
- United States (94):
  - Teva Investigational Site 13628, Birmingham, Alabama
  - Teva Investigational Site 13577, Birmingham, Alabama
  - Teva Investigational Site 13606, Phoenix, Arizona
  - Teva Investigational Site 13579, Phoenix, Arizona
  - Teva Investigational Site 13602, Little Rock, Arkansas
  - Teva Investigational Site 13568, Encino, California
  - Teva Investigational Site 13546, Fullerton, California
  - Teva Investigational Site 13540, Long Beach, California
  - Teva Investigational Site 13632, Redlands, California
  - Teva Investigational Site 13571, Redondo Beach, California
  - Teva Investigational Site 13573, San Diego, California
  - Teva Investigational Site 13538, Santa Monica, California
  - Teva Investigational Site 13594, Santa Rosa, California
  - Teva Investigational Site 13595, Walnut Creek, California
  - Teva Investigational Site 13629, Aurora, Colorado
  - Teva Investigational Site 13557, Boulder, Colorado
  - Teva Investigational Site 13593, Colorado Springs, Colorado
  - Teva Investigational Site 13633, Denver, Colorado
  - Teva Investigational Site 13612, Denver, Colorado
  - Teva Investigational Site 13631, Englewood, Colorado
  - Teva Investigational Site 13563, East Hartford, Connecticut
  - Teva Investigational Site 13550, Stamford, Connecticut
  - Teva Investigational Site 13635, Bradenton, Florida
  - Teva Investigational Site 13597, Gainesville, Florida
  - Teva Investigational Site 13607, Hialeah, Florida
  - Teva Investigational Site 13559, Jacksonville, Florida
  - Teva Investigational Site 13584, Ocala, Florida
  - Teva Investigational Site 13587, Orlando, Florida
  - Teva Investigational Site 13551, Orlando, Florida
  - Teva Investigational Site 13555, Orlando, Florida
  - Teva Investigational Site 13599, Orlando, Florida
  - Teva Investigational Site 13553, Pembroke Pines, Florida
  - Teva Investigational Site 13616, Pinellas Park, Florida
  - Teva Investigational Site 13567, West Palm Beach, Florida
  - Teva Investigational Site 13620, Atlanta, Georgia
  - Teva Investigational Site 13537, Atlanta, Georgia
  - Teva Investigational Site 13604, Boise, Idaho
  - Teva Investigational Site 13604, Meridian, Idaho
  - Teva Investigational Site 13585, Chicago, Illinois
  - Teva Investigational Site 13621, Chicago, Illinois
  - Teva Investigational Site 13627, Evanston, Illinois
  - Teva Investigational Site 13596, Indianapolis, Indiana
  - Teva Investigational Site 13617, Wichita, Kansas
  - Teva Investigational Site 13598, Wichita, Kansas
  - Teva Investigational Site 13566, Louisville, Kentucky
  - Teva Investigational Site 13603, Metairie, Louisiana
  - Teva Investigational Site 13582, Baltimore, Maryland
  - Teva Investigational Site 13582, Pikesville, Maryland
  - Teva Investigational Site 13590, Boston, Massachusetts
  - Teva Investigational Site 13589, New Bedford, Massachusetts
  - Teva Investigational Site 13543, Wellesley Hills, Massachusetts
  - Teva Investigational Site 13539, Ann Arbor, Michigan
  - Teva Investigational Site 13542, Golden Valley, Minnesota
  - Teva Investigational Site 13534, Kansas City, Missouri
  - Teva Investigational Site 13536, Springfield, Missouri
  - Teva Investigational Site 13619, St Louis, Missouri
  - Teva Investigational Site 13618, Fremont, Nebraska
  - Teva Investigational Site 13605, Las Vegas, Nevada
  - Teva Investigational Site 13578, Lebanon, New Hampshire
  - Teva Investigational Site 13575, Martinsville, New Jersey
  - Teva Investigational Site 13575, Raritan, New Jersey
  - Teva Investigational Site 13588, Albuquerque, New Mexico
  - Teva Investigational Site 13576, Amherst, New York
  - Teva Investigational Site 13565, Plainview, New York
  - Teva Investigational Site 13544, Greensboro, North Carolina
  - Teva Investigational Site 13574, Greensboro, North Carolina
  - Teva Investigational Site 13545, Raleigh, North Carolina
  - Teva Investigational Site 13609, Akron, Ohio
  - Teva Investigational Site 13634, Akron, Ohio
  - Teva Investigational Site 13533, Cincinnati, Ohio
  - Teva Investigational Site 13624, Cincinnati, Ohio
  - Teva Investigational Site 13569, Cleveland, Ohio
  - Teva Investigational Site 13626, Columbus, Ohio
  - Teva Investigational Site 13625, Mogadore, Ohio
  - Teva Investigational Site 13561, Oklahoma City, Oklahoma
  - Teva Investigational Site 13601, Eugene, Oregon
  - Teva Investigational Site 13591, Jenkintown, Pennsylvania
  - Teva Investigational Site 13554, Philadelphia, Pennsylvania
  - Teva Investigational Site 13608, Uniontown, Pennsylvania
  - Teva Investigational Site 13615, Greer, South Carolina
  - Teva Investigational Site 13556, Mt. Pleasant, South Carolina
  - Teva Investigational Site 13560, Bristol, Tennessee
  - Teva Investigational Site 13532, Nashville, Tennessee
  - Teva Investigational Site 13552, Nashville, Tennessee
  - Teva Investigational Site 13541, Austin, Texas
  - Teva Investigational Site 13623, Dallas, Texas
  - Teva Investigational Site 13611, Plano, Texas
  - Teva Investigational Site 13572, San Antonio, Texas
  - Teva Investigational Site 13614, Murray, Utah
  - Teva Investigational Site 13581, West Jordan, Utah
  - Teva Investigational Site 13630, Virginia Beach, Virginia
  - Teva Investigational Site 13564, Seattle, Washington
  - Teva Investigational Site 13586, Seattle, Washington
  - Teva Investigational Site 13600, Morgantown, West Virginia
- Canada (5):
  - Teva Investigational Site 11124, Hamilton, Ontario
  - Teva Investigational Site 11120, Calgary
  - Teva Investigational Site 11121, Montreal
  - Teva Investigational Site 11122, Newmarket
  - Teva Investigational Site 11123, Sarnia
- Czechia (7):
  - Teva Investigational Site 54144, Brno
  - Teva Investigational Site 54141, Kunratice
  - Teva Investigational Site 54145, Pardubice
  - Teva Investigational Site 54143, Prague
  - Teva Investigational Site 54146, Prague
  - Teva Investigational Site 54142, Prague
  - Teva Investigational Site 54142, Prague-4-Krc
- Finland (3):
  - Teva Investigational Site 40018, Helsinki
  - Teva Investigational Site 40017, Helsinki
  - Teva Investigational Site 40016, Turku
- Israel (6):
  - Teva Investigational Site 80096, Holon
  - Teva Investigational Site 80099, Jerusalem
  - Teva Investigational Site 80098, Nahariya
  - Teva Investigational Site 80097, Netanya
  - Teva Investigational Site 80100, Ramat Gan
  - Teva Investigational Site 80095, Tel Aviv
- Japan (19):
  - Teva Investigational Site 84072, Chofu-shi
  - Teva Investigational Site 84064, Chofu-shi
  - Teva Investigational Site 84066, Kagoshima
  - Teva Investigational Site 84069, Kai
  - Teva Investigational Site 84069, Kaisho
  - Teva Investigational Site 84073, Kawasaki
  - Teva Investigational Site 84073, Kawasaki-shi
  - Teva Investigational Site 84067, Kyoto
  - Teva Investigational Site 84062, Osaka
  - Teva Investigational Site 84070, Saitama
  - Teva Investigational Site 84070, Saitama-shi
  - Teva Investigational Site 84061, Sendai
  - Teva Investigational Site 84065, Shimotsuma
  - Teva Investigational Site 84063, Shinjuku-ku
  - Teva Investigational Site 84068, Shizuoka
  - Teva Investigational Site 84065, Tochigi
  - Teva Investigational Site 84064, Tokyo
  - Teva Investigational Site 84071, Toyonaka
  - Teva Investigational Site 84071, Toyonaka-shi
- Poland (5):
  - Teva Investigational Site 53364, Krakow
  - Teva Investigational Site 53363, Krakow
  - Teva Investigational Site 53366, Lublin
  - Teva Investigational Site 53365, Poznan
  - Teva Investigational Site 53367, Warsaw
- Russia (7):
  - Teva Investigational Site 50399, Kazan'
  - Teva Investigational Site 50395, Kazan'
  - Teva Investigational Site 50394, Moscow
  - Teva Investigational Site 50400, Moscow
  - Teva Investigational Site 50398, Nizhny Novgorod
  - Teva Investigational Site 50396, Nizhny Novgorod
  - Teva Investigational Site 50397, Ufa
- Spain (4):
  - Teva Investigational Site 31207, Madrid
  - Teva Investigational Site 31208, Pamplona
  - Teva Investigational Site 31205, Valladolid
  - Teva Investigational Site 31206, Zaragoza

REFERENCES:
- [Derived] McAllister P, Cohen JM, Campos VR, Ning X, Janka L, Barash S. Impact of fremanezumab on disability outcomes in patients with episodic and chronic migraine: a pooled analysis of phase 3 studies. J Headache Pain. 2022 Aug 29;23(1):112. doi: 10.1186/s10194-022-01438-4. PMID 36038833
- [Derived] Diener HC, McAllister P, Jurgens TP, Kessler Y, Ning X, Cohen JM, Campos VR, Barash S, Silberstein SD. Safety and tolerability of fremanezumab in patients with episodic and chronic migraine: a pooled analysis of phase 3 studies. Cephalalgia. 2022 Jul;42(8):769-780. doi: 10.1177/03331024221076485. Epub 2022 Mar 25. PMID 35331009
- [Derived] Nahas SJ, Naegel S, Cohen JM, Ning X, Janka L, Campos VR, Krasenbaum LJ, Holle-Lee D, Kudrow D, Lampl C. Efficacy and safety of fremanezumab in clinical trial participants aged >/=60 years with episodic or chronic migraine: pooled results from 3 randomized, double-blind, placebo-controlled phase 3 studies. J Headache Pain. 2021 Nov 24;22(1):141. doi: 10.1186/s10194-021-01351-2. PMID 34819017
- [Derived] Silberstein SD, Cohen JM, Yang R, Gandhi SK, Du E, Jann AE, Marmura MJ. Treatment benefit among migraine patients taking fremanezumab: results from a post hoc responder analysis of two placebo-controlled trials. J Headache Pain. 2021 Jan 7;22(1):2. doi: 10.1186/s10194-020-01212-4. PMID 33413075
- [Derived] Brandes JL, Kudrow D, Yeung PP, Sakai F, Aycardi E, Blankenbiller T, Grozinski-Wolff M, Yang R, Ma Y. Effects of fremanezumab on the use of acute headache medication and associated symptoms of migraine in patients with episodic migraine. Cephalalgia. 2020 Apr;40(5):470-477. doi: 10.1177/0333102419885905. Epub 2019 Nov 21. PMID 31752521
- [Derived] Dodick DW, Silberstein SD, Bigal ME, Yeung PP, Goadsby PJ, Blankenbiller T, Grozinski-Wolff M, Yang R, Ma Y, Aycardi E. Effect of Fremanezumab Compared With Placebo for Prevention of Episodic Migraine: A Randomized Clinical Trial. JAMA. 2018 May 15;319(19):1999-2008. doi: 10.1001/jama.2018.4853. PMID 29800211

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 2995 patients with migraine provided written informed consent. Of the 2995 patients screened, 875 met entry criteria, including diagnostic criteria for episodic migraine (EM) and diary compliance during the run-in period, and were randomized into this study from 123 study centers by 123 investigators.
Groups:
- Placebo: Participants randomized to receive placebo received three 1.5-mL placebo injections on Day 0, and a single 1.5-mL placebo injection on Days 28 and 56.
Period: Overall Study
Arm/Group | Placebo | Fremanezumab 675 mg/Placebo/Placebo | Fremanezumab 225/225/225 mg
Started | 294 | 291 | 290
Intent to Treat (ITT) | 294 | 291 | 290
Safety Population | 294 | 291 | 289
Full Analysis Set | 290 | 288 | 287
Completed | 265 | 264 | 262
Not Completed | 29 | 27 | 28
Not completed — Adverse Event | 7 | 5 | 4
Not completed — Withdrawal by Subject | 5 | 8 | 13
Not completed — Protocol Violation | 2 | 3 | 7
Not completed — Lost to Follow-up | 12 | 9 | 4
Not completed — Other | 1 | 1 | 0
Not completed — Pregnancy | 2 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intent to treat (ITT) population
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Fremanezumab 675 mg/Placebo/Placebo | Fremanezumab 225/225/225 mg | Total
Number analyzed (Participants) | 294 | 291 | 290 | 875
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.3 (12.04) | 41.1 (11.41) | 42.9 (12.67) | 41.8 (12.06)
Age, Customized [Count of Participants; unit: Participants]
  18-45 years | 184 | 178 | 163 | 525
  46-65 years | 102 | 110 | 120 | 332
  >65 years | 8 | 3 | 7 | 18
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 247 | 251 | 244 | 742
  Male | 47 | 40 | 46 | 133
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 225 | 232 | 243 | 700
  Black | 40 | 28 | 18 | 86
  Asian | 25 | 27 | 25 | 77
  American Indian or Alaska Native | 0 | 1 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Other | 4 | 2 | 1 | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Not Hispanic or Latino | 267 | 251 | 252 | 770
  Hispanic or Latino | 27 | 39 | 37 | 103
  Unknown | 0 | 1 | 1 | 2
Preventive Medication Use During Baseline Period [Count of Participants; unit: Participants] — Eligible patients entered a 28-day run-in/baseline period during which headache information was captured daily throughout study participation using the electronic headache diary device. During randomization, patients were stratified based on sex, country, and baseline preventive migraine medication use (yes, no) to ensure balance for the covariates.
  Participants
    Yes | 62 | 58 | 62 | 182
    No | 232 | 233 | 228 | 693
Weight [Mean (Standard Deviation); unit: kg] | 75.3 (16.01) | 74.2 (15.42) | 72.1 (15.77) | 73.9 (15.77)
Time Since Initial Migraine Diagnosis [Mean (Standard Deviation); unit: years] | 19.9 (11.87) | 20.0 (12.14) | 20.7 (12.85) | 20.2 (12.28)
Total Number of Headache Days of Any Duration And Any Severity During the 28 Day Baseline Period [Mean (Standard Deviation); unit: days] — Eligible patients entered a 28-day run-in/baseline period during which headache information was captured daily throughout study participation using the electronic headache diary device. Population: Three participants did not capture data in the e-diary.
  days
    number analyzed (Participants) | 293 | 291 | 288 | 872
    (all) | 11.2 (2.45) | 11.1 (2.42) | 11.0 (2.49) | 11.1 (2.45)
Number of Migraine Days [Mean (Standard Deviation); unit: days] — Eligible patients entered a 28-day run-in/baseline period during which headache information was captured daily throughout study participation using the electronic headache diary device. Migraine headaches are as defined in The International Classification of Headache Disorders 3rd edition (ICHD-3). Population: Three participants did not capture data in the e-diary.
  days
    number analyzed (Participants) | 293 | 291 | 288 | 872
    (all) | 9.1 (2.65) | 9.3 (2.65) | 8.9 (2.63) | 9.1 (2.64)
Number of Headache Days of At Least Moderate Severity [Mean (Standard Deviation); unit: days] — Eligible patients entered a 28-day run-in/baseline period during which headache information was captured daily throughout study participation using the electronic headache diary device. Headache severity was subjectively rated by the patient as mild, moderate or severe. Population: Three participants did not capture data in the e-diary.
  days
    number analyzed (Participants) | 293 | 291 | 288 | 872
    (all) | 6.9 (3.12) | 7.2 (3.14) | 6.8 (2.90) | 7.0 (3.06)
Number of Days of Use of Any Acute Headache Medications [Mean (Standard Deviation); unit: days] — Eligible patients entered a 28-day run-in/baseline period during which headache information (including information about use of headache medications) was captured daily throughout study participation using the electronic headache diary device. Population: Three participants did not capture data in the e-diary.
  days
    number analyzed (Participants) | 293 | 291 | 288 | 872
    (all) | 7.7 (3.60) | 7.8 (3.74) | 7.7 (3.37) | 7.8 (3.57)
Migraine Disability Assessment (MIDAS) Total Score [Mean (Standard Deviation); unit: units on a scale] — The MIDAS questionnaire is a 5-item instrument developed to assess headache-related disability based on lost days of activity in 3 domains (work, household work, and nonwork) over the previous 3 months. The total score, ie, the sum of the # lost days answered for the first 5 questions, is used for grading of disability, with scores of 0-5 = grade 1 (little or no disability), 6-10 =grade 2 (mild disability), 11-20 = grade 3 (moderate disability), and ≥21 interpreted as grade 4 (severe disability). Population: Eleven participants did not capture data in the e-diary.
  units on a scale
    number analyzed (Participants) | 290 | 287 | 287 | 864
    (all) | 37.3 (27.59) | 41.7 (32.96) | 38.0 (33.19) | 39.0 (31.36)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Monthly Average Number of Migraine Days During the 12-Week Period After the First Dose of Study Drug
Description: A migraine day was defined as when at least 1 of the following situations occurred: - a calendar day (0:00 to 23:59) demonstrating at least 4 consecutive hours of a headache endorsing criteria for migraine with or without aura - a calendar day (0:00 to 23:59) demonstrating at least 4 consecutive hours of a headache endorsing criteria for probable migraine, a migraine subtype where only 1 migraine criterion is missing - a calendar day (0:00 to 23:59) demonstrating a headache of any duration that was treated with migraine-specific medications (triptans and ergot compounds) Monthly averages are derived and normalized to 28 days equivalent by the following formula: (# days of efficacy variable over relevant period / # days with assessments recorded in the e-diary over the relevant period) * 28. The change is calculated as postbaseline value - baseline value.
Time Frame: Baseline (Days -28 to Day -1), Treatment (Days 1 - Week 12)
Population: Full analysis set
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Placebo | Fremanezumab 675 mg/Placebo/Placebo | Fremanezumab 225/225/225 mg
Number analyzed (Participants) | 290 | 288 | 287
days | -2.7 [-4.7 to -0.5] | -4.0 [-6.4 to -1.9] | -4.2 [-6.2 to -2.0]
Statistical Analysis 1: Comparison: Placebo vs Fremanezumab 675 mg/Placebo/Placebo; Due to the deviation from the normal distribution assumption of the data, the primary analysis was conducted using the Wilcoxon rank-sum test as outlined in the SAP; Test type: Superiority; p < 0.0001, Wilcoxon (Mann-Whitney) — 0.05 level of significance
Statistical Analysis 2: Comparison: Placebo vs Fremanezumab 225/225/225 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, Wilcoxon (Mann-Whitney) — 0.05 level of significance

2. Primary Outcome: Participants With Adverse Events
Description: An adverse event was defined as any untoward medical occurrence that develops or worsens in severity during the conduct of a clinical study and does not necessarily have a causal relationship to the study drug. Severity was rated by the investigator on a scale of mild, moderate and severe, with severe= an AE which prevents usual activities. Relationship of AE to treatment was determined by the investigator. Serious AEs include death, a life-threatening adverse event, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, OR an important medical event that jeopardized the patient and required medical intervention to prevent the previously listed serious outcomes.
Time Frame: Day 1 to Week 12
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Fremanezumab 675 mg/Placebo/Placebo | Fremanezumab 225/225/225 mg
Number analyzed (Participants) | 293 | 291 | 290
Participants
  Any AEs | 171 | 193 | 192
  Severe AEs | 11 | 16 | 10
  Treatment-related AEs | 109 | 137 | 138
  Serious adverse events | 7 | 3 | 3
  Deaths | 0 | 1 | 0
  Discontinued from study due to AE | 5 | 5 | 5

3. Secondary Outcome: Percentage of Participants With At Least 50% Reduction In Monthly Average Number of Migraine Days During the 12-Week Period After the First Dose of Study Drug
Description: Responder rates were defined as the percentage of total subjects who reached at least a 50% reduction in the monthly average of headache days (as subjectively reported by participants in the study diary) of at least moderate severity relative to the baseline period. For the overall analysis (Month 1-3), patients who discontinued early were considered nonresponders. Monthly averages are derived and normalized to 28 days equivalent by the following formula: (# days of efficacy variable over relevant period / # days with assessments recorded in the e-diary over the relevant period) * 28. The percentage reduction in monthly average is calculated as: ((baseline value - postbaseline value) / baseline value) * 100
Time Frame: Baseline (Days -28 to Day -1), Treatment Month 1, Month 2, Month 3, Month 1-3 (Days 1 - Week 12)
Population: Full analysis set
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Fremanezumab 675 mg/Placebo/Placebo | Fremanezumab 225/225/225 mg
Number analyzed (Participants) | 290 | 288 | 287
percentage of participants
  Month 1 | 25.2 | 44.1 | 47.0
  Month 2: number analyzed (Participants) | 274 | 274 | 274
  Month 2 | 34.8 | 46.9 | 48.4
  Month 3: number analyzed (Participants) | 268 | 269 | 263
  Month 3 | 37.2 | 49.0 | 51.2
  Overall - Months 1-3 | 27.9 | 44.4 | 47.7
Statistical Analysis 1: Comparison: Placebo vs Fremanezumab 675 mg/Placebo/Placebo; Month 1 P-value based on Cochran-Mantel-Haenszel test stratified by baseline preventive medication use; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — 0.05 level of significance
Statistical Analysis 2: Comparison: Placebo vs Fremanezumab 225/225/225 mg; Month 1 P-value based on Cochran-Mantel-Haenszel test stratified by baseline preventive medication use; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — 0.05 level of significance
Statistical Analysis 3: Comparison: Placebo vs Fremanezumab 675 mg/Placebo/Placebo; Month 2 P-value based on Cochran-Mantel-Haenszel test stratified by baseline preventive medication use; Test type: Superiority; p = 0.0032, Cochran-Mantel-Haenszel — 0.05 level of significance
Statistical Analysis 4: Comparison: Placebo vs Fremanezumab 225/225/225 mg; Month 2 P-value based on Cochran-Mantel-Haenszel test stratified by baseline preventive medication use; Test type: Superiority; p = 0.0010, Cochran-Mantel-Haenszel — 0.05 level of significance
Statistical Analysis 5: Comparison: Placebo vs Fremanezumab 675 mg/Placebo/Placebo; Month 3 P-value based on Cochran-Mantel-Haenszel test stratified by baseline preventive medication use; Test type: Superiority; p = 0.0048, Cochran-Mantel-Haenszel — 0.05 level of significance
Statistical Analysis 6: Comparison: Placebo vs Fremanezumab 225/225/225 mg; Month 3 P-value based on Cochran-Mantel-Haenszel test stratified by baseline preventive medication use; Test type: Superiority; p = 0.0003, Cochran-Mantel-Haenszel — 0.05 level of significance
Statistical Analysis 7: Comparison: Placebo vs Fremanezumab 675 mg/Placebo/Placebo; Overall P-value based on Cochran-Mantel-Haenszel test stratified by baseline preventive medication use; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — 0.05 level of significance
Statistical Analysis 8: Comparison: Placebo vs Fremanezumab 225/225/225 mg; Overall P-value based on Cochran-Mantel-Haenszel test stratified by baseline preventive medication use; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — 0.05 level of significance

4. Secondary Outcome: Change From Baseline in the Monthly Average Number of Days of Use of Any Acute Headache Medicine During the 12 Week Period After the First Dose of Study Drug
Description: Patients recorded any migraine medications (name of drug, number of tablets/capsules, and the dose in milligrams per tablet/capsule) taken on each day in their electronic headache diary device. Acute migraine-specific medication included triptans or ergots. Monthly averages are derived and normalized to 28 days equivalent by the following formula: (# days of efficacy variable over relevant period / # days with assessments recorded in the e-diary over the relevant period) * 28. The change is calculated as postbaseline value - baseline value.
Time Frame: Baseline (Days -28 to Day -1), Treatment (Days 1 - Week 12)
Population: Full analysis set
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Placebo | Fremanezumab 675 mg/Placebo/Placebo | Fremanezumab 225/225/225 mg
Number analyzed (Participants) | 290 | 288 | 287
days | -1.7 [-4.0 to 0.0] | -3.0 [-5.6 to -0.8] | -3.2 [-5.2 to -1.2]
Statistical Analysis 1: Comparison: Placebo vs Fremanezumab 675 mg/Placebo/Placebo; Due to the deviation from the normal distribution assumption of the data, the Wilcoxon rank-sum test was conducted as the primary analysis for each active treatment group and placebo treatment group for this endpoint; Test type: Superiority; p < 0.0001, Wilcoxon (Mann-Whitney) — 0.05 level of significance
Statistical Analysis 2: Comparison: Placebo vs Fremanezumab 225/225/225 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p < 0.0001, Wilcoxon (Mann-Whitney) — 0.05 level of significance

5. Secondary Outcome: Change From Baseline in the Number of Migraine Days During the 4 Week Period After the First Dose of Study Drug
Description: as for outcome 1
Time Frame: Baseline (Days -28 to Day -1), Treatment (Days 1 - Week 4)
Population: Full analysis set; includes participants with observations
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Placebo | Fremanezumab 675 mg/Placebo/Placebo | Fremanezumab 225/225/225 mg
Number analyzed (Participants) | 290 | 285 | 286
days | -2.0 [-4.2 to 0.5] | -4.0 [-6.2 to -1.3] | -4.0 [-6.1 to -1.7]
Statistical Analysis 1: Comparison: Placebo vs Fremanezumab 675 mg/Placebo/Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p < 0.0001, Wilcoxon (Mann-Whitney) — 0.05 level of significance
Statistical Analysis 2: Comparison: Placebo vs Fremanezumab 225/225/225 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p < 0.0001, Wilcoxon (Mann-Whitney) — 0.05 level of significance

6. Secondary Outcome: Change From Baseline in the Monthly Average Number of Migraine Days During the 12 Week Period After the First Dose of Study Medication in Patients Not Receiving Concomitant Preventive Migraine Medications
Description: A subset of patients (specified in the protocol not to exceed 30%) were allowed to use 1 concomitant migraine preventive medication. This outcome only includes those participants who did not take concomitant preventive migraine medication during this study. A migraine day has been previously defined. Monthly averages are derived and normalized to 28 days equivalent by the following formula: (# days of efficacy variable over relevant period / # days with assessments recorded in the e-diary over the relevant period) * 28. The change is calculated as postbaseline value - baseline value.
Time Frame: Baseline (Days -28 to Day -1), Treatment (Days 1 - Week 12)
Population: Full analysis set of participants who did not receive concomitant migraine prevention medication
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Placebo | Fremanezumab 675 mg/Placebo/Placebo | Fremanezumab 225/225/225 mg
Number analyzed (Participants) | 230 | 230 | 225
days | -2.9 [-4.9 to -0.6] | -4.0 [-6.3 to -2.0] | -4.2 [-6.2 to -2.0]
Statistical Analysis 1: Comparison: Placebo vs Fremanezumab 675 mg/Placebo/Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p < 0.0001, Wilcoxon (Mann-Whitney) — 0.05 level of significance
Statistical Analysis 2: Comparison: Placebo vs Fremanezumab 225/225/225 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p < 0.0001, Wilcoxon (Mann-Whitney) — 0.05 level of significance

7. Secondary Outcome: Change From Baseline in Migraine-Related Disability Score (MIDAS), As Measured by the Migraine Disability Assessment At 4 Weeks After the Last (3rd) Dose of Study Drug
Description: The MIDAS questionnaire is a 5-item instrument developed to assess headache-related disability based on lost days of activity in 3 domains (work, household work, and nonwork) over the previous 3 months. The total score, ie, the sum of the # lost days answered for the first 5 questions, is used for grading of disability, with scores of 0-5 lost days = grade 1 (little or no disability), 6-10 lost days =grade 2 (mild disability), 11-20 lost days = grade 3 (moderate disability), and ≥21 lost days interpreted as grade 4 (severe disability). Negative change from baseline scores indicate a reduction (improvement) in headache-related disability.
Time Frame: Baseline (Day 0), Treatment Week 12 (4 weeks after the 3rd dose)
Population: Full analysis set
Measure: Median (Inter-Quartile Range); unit: lost days
Arm/Group | Placebo | Fremanezumab 675 mg/Placebo/Placebo | Fremanezumab 225/225/225 mg
Number analyzed (Participants) | 290 | 288 | 287
lost days | -12.5 [-29.5 to -2.0] | -18.0 [-39.0 to -6.0] | -19.0 [-36.0 to -7.0]
Statistical Analysis 1: Comparison: Placebo vs Fremanezumab 675 mg/Placebo/Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.0023, Wilcoxon (Mann-Whitney) — 0.05 level of significance
Statistical Analysis 2: Comparison: Placebo vs Fremanezumab 225/225/225 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.0021, Wilcoxon (Mann-Whitney) — 0.05 level of significance

8. Secondary Outcome: Electrocardiogram Finding Shifts From Baseline to Overall
Description: 12-lead ECGs were performed before other assessments (eg, blood draws and administration of questionnaires) and performed in triplicate. The worst post-baseline finding for the patient is summarized. Only patients with both baseline and post-baseline ECGs are included. The ECG was evaluated by the investigator at the time of recording (signed and dated), and the printout was kept in the source documentation file. When potentially clinically significant findings were detected by the investigator, a cardiologist at a central diagnostic center was consulted for a definitive interpretation. Any ECG finding that was judged by the investigator as a potentially clinically significant change (worsening) compared with a baseline value was considered an adverse event. - NCS = abnormal, not clinically significant - CS = abnormal, clinically significant Shift format is: baseline finding / worst post-baseline finding
Time Frame: Baseline (Day 0), Treatment Week 12 (or early withdrawal)
Population: Safety population of participants with both baseline and post-treatment ECGs
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Fremanezumab 675 mg/Placebo/Placebo | Fremanezumab 225/225/225 mg
Number analyzed (Participants) | 278 | 276 | 281
Participants
  Normal / Normal | 161 | 169 | 181
  Normal / NCS | 32 | 41 | 25
  Normal / CS | 0 | 0 | 0
  NCS / Normal | 27 | 23 | 29
  NCS / NCS | 58 | 43 | 46
  NCS / CS | 0 | 0 | 0
  CS / Normal | 0 | 0 | 0
  CS / NCS | 0 | 0 | 0
  CS / CS | 0 | 0 | 0

9. Secondary Outcome: Participants With Vital Signs Potentially Clinically Significant Abnormal Values
Description: Vital signs were performed before other assessments (eg, blood draws and administration of questionnaires). Vital signs with at least one participant showing potentially clinically significant abnormal findings included: - Pulse Rate Low: <=50 and decrease of >=15 beats per minute - Systolic Blood Pressure Low: <=90 mmHg and decrease of >=20 mmHg - Diastolic Blood Pressure High: >=105 mmHg and increase of >=15 mmHg - Diastolic Blood Pressure Low: <=50 mmHg and decrease of >=15 mmHg - Respiratory Rate Low: <10 breaths / minute
Time Frame: Treatment Days 28, 56 and 84. Changes from previous reading may reflect the baseline reading performed on Day 0.
Population: Safety population of participants with both baseline and post-treatment values for each vital sign.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Fremanezumab 675 mg/Placebo/Placebo | Fremanezumab 225/225/225 mg
Number analyzed (Participants) | 285 | 285 | 285
Participants
  Participants with at least 1 abnormality | 3 | 4 | 5
  Pulse Rate Low | 0 | 1 | 0
  Systolic Blood Pressure Low | 0 | 2 | 1
  Diastolic Blood Pressure High | 0 | 1 | 2
  Diastolic Blood Pressure Low | 2 | 1 | 0
  Respiratory Rate Low | 1 | 0 | 2

10. Secondary Outcome: Participants With Serum Chemistry and Hematology Potentially Clinically Significant Abnormal Results
Description: Serum chemistry and hematology laboratory tests with potentially clinically significant abnormal findings included: - Blood Urea Nitrogen (BUN) High: >=10.71 mmol/L - Bilirubin High: >=34.2 umol/L - Alanine Aminotransferase (ALT): >=3*upper limit of normal (ULN) - Aspartate Aminotransferase (AST): >=3*upper limit of normal (ULN) - Gamma Glutamyl Transferase (GGT): >=3*upper limit of normal (ULN) - Hemoglobin: Male: <115 g/L or Female: <=95 g/L - Hematocrit: Male: <0.37 L/L or Female: <0.32 L/L - Leukocytes: >=20*10^9/L or <=3*10^9/L - Eosinophils/Leukocytes: >=10% - Platelets: >=700*10^9/L or <=75*10^9/L
Time Frame: Treatment Days 28, 56 and 84 (or early withdrawal)
Population: Safety population of participants with at least one postbaseline result for the tests.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Fremanezumab 675 mg/Placebo/Placebo | Fremanezumab 225/225/225 mg
Number analyzed (Participants) | 285 | 285 | 285
Participants
  Blood Urea Nitrogen (BUN) | 1 | 0 | 1
  Bilirubin | 1 | 0 | 1
  Alanine Aminotransferase (ALT) | 0 | 1 | 0
  Aspartate Aminotransferase (AST) | 0 | 0 | 1
  Gamma Glutamyl Transferase (GGT) | 4 | 4 | 8
  Hemoglobin | 1 | 4 | 2
  Hematocrit | 3 | 6 | 6
  Leukocytes | 4 | 1 | 6
  Eosinophils/Leukocytes | 7 | 3 | 5
  Platelets | 1 | 0 | 0

11. Secondary Outcome: Participants With Urinalysis Laboratory Tests Potentially Clinically Significant Abnormal Results
Description: Urinalysis with potentially clinically significant abnormal findings included: - Blood: >=2 unit increase from baseline - Urine Glucose (mg/dL): >=2 unit increase from baseline - Ketones (mg/dL): >=2 unit increase from baseline - Urine Protein (mg/dL): >=2 unit increase from baseline
Time Frame: Treatment Days 28, 56 and 84. Changes from previous reading reflect the baseline reading performed on Day 0.
Population: Safety population of participants with at least one postbaseline result for the tests
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Fremanezumab 675 mg/Placebo/Placebo | Fremanezumab 225/225/225 mg
Number analyzed (Participants) | 285 | 285 | 285
Participants
  Participants with at least 1 abnormality | 55 | 54 | 49
  Blood | 29 | 30 | 23
  Urine glucose | 5 | 8 | 2
  Ketones | 5 | 7 | 9
  Urine protein | 25 | 19 | 23

12. Secondary Outcome: Prothrombin Time Shifts From Baseline to Endpoint
Description: Shifts in prothrombin time from baseline to endpoint were summarized using patient counts grouped into three categories: - Low (below normal range) - Normal (within the normal range of 9.4 to 12.5 seconds) - High (above normal range) Shift format is: baseline finding / endpoint finding
Time Frame: Baseline (Day 0), Treatment Endpoint (Week 12)
Population: Safety population of participants with both baseline and posttreatment values
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Fremanezumab 675 mg/Placebo/Placebo | Fremanezumab 225/225/225 mg
Number analyzed (Participants) | 284 | 285 | 284
Participants
  Low / Low | 0 | 0 | 0
  Low / Normal | 0 | 1 | 1
  Low / High | 0 | 0 | 0
  Normal / Low | 0 | 1 | 0
  Normal / Normal | 254 | 248 | 250
  Normal / High | 14 | 10 | 13
  High / Low | 0 | 0 | 0
  High / Normal | 8 | 15 | 12
  High / High | 8 | 10 | 8

13. Secondary Outcome: Injection Site Reaction Adverse Events
Description: Counts of participants who reported treatment-emergent injection site reactions as AEs are summarized. Preferred terms from MedDRA version 18.1 are offered without a threshold applied.
Time Frame: Day 1 to Week 12
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Fremanezumab 675 mg/Placebo/Placebo | Fremanezumab 225/225/225 mg
Number analyzed (Participants) | 293 | 291 | 290
Participants
  Participants with >=1 injection site reaction | 106 | 131 | 130
  Injection site pain | 76 | 86 | 87
  Injection site induration | 45 | 57 | 71
  Injection site erythema | 41 | 55 | 52
  Injection site haemorrhage | 6 | 9 | 3
  Injection site pruritus | 2 | 4 | 4
  Injection site swelling | 0 | 2 | 3
  Injection site urticaria | 2 | 2 | 1
  Injection site rash | 0 | 1 | 3
  Fatigue | 0 | 1 | 0
  Injection site bruising | 1 | 0 | 0
  Injection site dermatitis | 0 | 0 | 1
  Injection site hypersensitivity | 0 | 0 | 1
  Injection site nodule | 0 | 0 | 1
  Injection site oedema | 0 | 0 | 1
  Injection site warmth | 0 | 1 | 0

14. Secondary Outcome: Participants With Positive Electronic Columbia Suicide Severity Rating Scale Results After the First Dose of Study Drug
Description: The electronic Columbia-Suicide Severity Rating Scale (eC-SSRS) was used to assess the patient's suicidal ideation (severity and intensity) and behavior (Posner et al 2011). The eC-SSRS Baseline/Screening version was completed by the patient at visit 2, and the eC-SSRS Since Last Visit version was completed by the patient at all other time points. Any positive findings on the eC-SSRS Since Last Visit version required evaluation by a physician or doctoral-level psychologist. Findings after the first dose of study drug using the eC-SSRS Since Last Visit version are summarized.
Time Frame: Day 1 to Week 12
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Fremanezumab 675 mg/Placebo/Placebo | Fremanezumab 225/225/225 mg
Number analyzed (Participants) | 294 | 291 | 289
Participants
  Suicidal Ideation | 0 | 0 | 2
  Suicidal Behaviour | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Day 1 to Week 12
Groups:
- Placebo: Participants randomized to receive placebo received three 1.5-mL placebo injections Day 0, and a single 1.5-mL placebo injection on Days 28 and 56.
- Fremanezumab 675 mg/Placebo/Placebo: Participants randomized to receive fremanezumab 675 mg/placebo/placebo received 675 mg of fremanezumab as 3 active injections (225 mg/1.5 mL) on Day 0, and placebo as a single 1.5-mL injection on Days 28 and 56.
Arm/Group | Placebo | Fremanezumab 225/225/225 mg | Fremanezumab 675 mg/Placebo/Placebo
All-Cause Mortality (participants affected / at risk) | 0/294 | 0/289 | 1/291
Serious Adverse Events (participants affected / at risk) | 7/294 | 3/289 | 3/291
Other Adverse Events (participants affected / at risk) | 113/294 | 132/289 | 133/291
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=294) | Fremanezumab 225/225/225 mg (N=289) | Fremanezumab 675 mg/Placebo/Placebo (N=291)
Intestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Death (General disorders) | 0 (0) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Tendon injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Lentigo maligna (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Generalised tonic-clonic seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Status migrainosus (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=294) | Fremanezumab 225/225/225 mg (N=289) | Fremanezumab 675 mg/Placebo/Placebo (N=291)
Injection site erythema (General disorders) | 41 (88) | 52 (102) | 55 (110)
Injection site induration (General disorders) | 45 (93) | 71 (134) | 57 (126)
Injection site pain (General disorders) | 76 (191) | 87 (245) | 86 (234)
Upper respiratory tract infection (Infections and infestations) | 15 (15) | 16 (17) | 11 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.

DOCUMENTS (2):
  • Study Protocol (2016-03-30): https://cdn.clinicaltrials.gov/large-docs/61/NCT02629861/Prot_000.pdf
  • Statistical Analysis Plan (2017-05-26): https://cdn.clinicaltrials.gov/large-docs/61/NCT02629861/SAP_001.pdf